CLINICAL TRIAL: NCT01195597
Title: Effect of an Electronic Nicotine Delivery Device (ENDD) on Smoking Cessation and Reduction: a Pilot Study
Brief Title: Smoking Cessation and Reduction With an Electronic Nicotine Delivery Device (ENDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Collaborators: Lega Italiana Anti Fumo (Other); Arbi Group Srl (Industry)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor of Internal Medicine, Universita degli Studi di Catania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT00/10
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Nicotine Dependence; Smoking Cessation
Keywords: electronic cigarette; ENDD; nicotine; smoking cessation; smoking reduction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Vaping; Smoking Reduction | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- E-Cigarette 7.2 mg nicotine (Experimental): Well characterized group of 40 regular smokers not intending to quit experimenting the E-Cigarette with 7.2 mg nicotine cartridges.
  Interventions: Device: E-Cigarette 7.2 mg nicotine

INTERVENTIONS:
Device: E-Cigarette 7.2 mg nicotine — Participants were given a free e-Cigarette kit containing two rechargeable batteries, a charger, and two atomizers and instructed on how to charge, activate and use the e-Cigarette. Key troubleshooting were addressed and phone numbers were supplied for both technical and medical assistance. A full 4-weeks supply of 7.2 mg nicotine cartridges ("Original" cartridges; Arbi Group Srl, Milano, Italy) was also provided and participants were trained on how to load them onto the e-Cigarette's atomizer
  Other Names: E-Cigarette with nicotine cartridges

SUMMARY:
The study's major aim is to investigate the ability of a commercial Electronic Nicotine Delivery Device (ENDD) to induce long-term smoking reduction/abstinence in smokers unwilling to quit. Secondary aims are to monitor adverse events and measure participants' perception and acceptance of the product.

This pilot study will evaluate smoking reduction/abstinence effects, product preferences, and adverse events of a currently marketed device in Italy ("Categoria" electronic cigarette - "ORIGINAL" 7.2 mg nicotine cartridges). The primary hypothesis is that the E-Cigarette is a safe device that allows smoking reduction or abstinence in smokers.

DETAILED DESCRIPTION:
Cigarette smoking continues to be a very difficult addiction to break. Therefore, improved approaches to smoking cessation are necessary. The electronic-cigarette (e-Cigarette), a battery-powered electronic nicotine delivery device (ENDD) resembling a cigarette, may help smokers to remain abstinent during their quit attempt or to reduce cigarette consumption. The efficacy of these devices in smoking cessation and/or smoking reduction studies has never been investigated.

In this prospective proof-of-concept study we monitored possible modifications in smoking habits of 40 smokers (unwilling to quit) experimenting the 'Categoria' e-Cigarette focusing on smoking reduction and smoking abstinence. Study participants were invited to attend four study visits: at baseline, week-4, week-8, and week-12. Product use, number of cigarettes smoked, and exhaled carbon monoxide (eCO) levels were measured at each visit. Smoking reduction and abstinence rates were calculated. Adverse events and product preferences were also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* healthy smokers
* unwilling to quit
* age 18-60 years
* smoking ≥ 15 cig/day for at least 5 years
* exhaled CO level of ≥ 15 ppm
* FTND ≥ 5

Exclusion Criteria:

* alcohol and illicit drug use
* breastfeeding or pregnancy
* major depression or other psychiatric conditions
* previous experience with ENDD
* recent myocardial infarction
* angina pectoris
* high blood pressure (BP>140mm Hg systolic and/or 90mmHg diastolic)
* diabetes mellitus
* severe allergies
* poorly controlled asthma or other airways diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Polosa, MD, PhD, Principal Investigator — Università di Catania
Locations (1):
- Dipartimento di Medicina Interna e Specialistica; Centro per la Prevenzione e Cura del Tabagismo (CPCT), Catania, Italy

REFERENCES:
- [Derived] Polosa R, Morjaria JB, Caponnetto P, Campagna D, Russo C, Alamo A, Amaradio M, Fisichella A. Effectiveness and tolerability of electronic cigarette in real-life: a 24-month prospective observational study. Intern Emerg Med. 2014 Aug;9(5):537-46. doi: 10.1007/s11739-013-0977-z. Epub 2013 Jul 20. PMID 23873169
- [Derived] Polosa R, Caponnetto P, Morjaria JB, Papale G, Campagna D, Russo C. Effect of an electronic nicotine delivery device (e-Cigarette) on smoking reduction and cessation: a prospective 6-month pilot study. BMC Public Health. 2011 Oct 11;11:786. doi: 10.1186/1471-2458-11-786. PMID 21989407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy smokers 18-60 years old, smoking ≥ 15 factorymade cigarettes per day (cig/day) for at least the past 10 years and not currently attempting to quit smoking or wishing to do so in the next 30 days were recruited, Italy. None of the participants reported a history of alcohol and drug use, major depression or other psychiatric conditions.
Groups:
- ENDD Group: Well characterized group of 40 regular smokers not intending to quit experimenting the E-Cigarette with 7.2 mg nicotine cartridges.
Period: Overall Study
Arm/Group | ENDD Group
Started | 40
Completed | 27
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | ENDD Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Region of Enrollment [Number; unit: participants]
  Italy | 40

OUTCOME MEASURES:

1. Primary Outcome: Sustained 50% Reduction in the Number of Cig/Day at Week-24 From Baseline (Reducers)
Description: Participants were monitored for up to 24 weeks. This is the number of smokers who sustained 50% reduction in the number of cig/day at week-24 from baseline (reducers).
Time Frame: number of cigarettes/day as assessed at week 24
Population: Intention to treat (ITT)
Measure: Number; unit: number of participants
Groups:
- Smokers Not Willing to Quit: 7.4 mg nicotine cartridges ("Original" cartridges; Arbi Group Srl, Milano, Italy)
Arm/Group | Smokers Not Willing to Quit
Number analyzed (Participants) | 40
number of participants | 13 [20 to 50]

2. Secondary Outcome: Sustained 80% Reduction in the Number of Cig/Day at Week- 24 From Baseline (Heavy Reducers)
Description: Participants were monitored for up to 24 weeks. This is the number of partecipants who sustained 80% reduction at week 24
Time Frame: number of cigarettes/day as assessed at week 24
Population: Intention to treat (ITT)
Measure: Number; unit: number of participants
Arm/Group | Smokers Not Willing to Quit
Number analyzed (Participants) | 40
number of participants | 5 [25 to 35]

ADVERSE EVENTS:
Time Frame: 6 months
Description: daily questionnaire
Arm/Group | ENDD Group
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 22/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENDD Group (N=40)
troat irritation (Skin and subcutaneous tissue disorders) | 11 (40)
mouth irritation (Skin and subcutaneous tissue disorders) | 11 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No